CLINICAL TRIAL: NCT06545318
Title: A Novel Sperm Selection Method Provides Advantages Over Conventional Approaches: Validation Through a Clinical Pilot Study
Brief Title: A Novel Sperm Selection Method Provides Advantages Over Conventional Approaches
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Center of Innovation Technology & Reproductive Medicine (Industry)
Collaborators: Universidad Nacional Autonoma de Mexico (Other)
Responsible Party: Principal Investigator, Liliana Berenice Ramírez Domínguez, Scientific Coordinator, Center of Innovation Technology & Reproductive Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: CI-21-101
Record Dates: First submitted 2024-07-22; First posted 2024-08-09 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Male Infertility
Keywords: Spem preparation; in vitro fertilization; Sperm membrane potential; Sperm intracellular calcium
MeSH Terms: conditions — Infertility, Male | interventions — Centrifugation, Density Gradient

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants did not know if their sperm would be selected by density gradient centrifugation ir the novel device (CA0 chamber)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Density Gradient Centrifugation (Active Comparator): A density gradient of is formed in 15 mL conical tubes as follows: 1 mL of lower gradient (90%) medium is placed at the bottom, 1 mL of upper (45%) gradient medium is placed on top of the bottom layer, and 1 mL of semen sample is layered above the gradient. Tubes are centrifuged for 10 minutes at 1,200 x g at room temperature. The pellet containing the viable cells is separated, resuspended in 1 mL of HTF-HEPES medium, and centrifuged at room temperature for 10 minutes at 1,200 x g to remove traces of gradient medium. The supernatant is then removed, 500 µL of HTF-HEPES medium are added to the sperm pellet, carefully mixed, and cells are counted
  Interventions: Device: Density Gradient Centrifugation
- CA0 chamber (Experimental): One mL of semen is placed in the base, then the intermediate part is placed on the base, taking care to match the notches that assemble both parts. Subsequently, 900 µL of HTF-HEPES medium are placed in the intermediate part, the cover is placed and the device is incubated at 37°C for 30 minutes. Subsequently, a 500-µL aliquot is recovered and cells are counted
  Interventions: Device: CA0 chamber

INTERVENTIONS:
Device: Density Gradient Centrifugation — Sperm separation with density gradients
  Arms: Density Gradient Centrifugation
Device: CA0 chamber — Sperm separation with a novel device
  Arms: CA0 chamber

SUMMARY:
The goal of this clinical trial is to know if a novel sperm selection device (CA0) has a similar performance than the standard selection method in teratozoospermic and azoospermic men. The main questions it aims to answer are:

Does the CA0 sperm selection device increases the sperm concentration? Does the CA0 sperm selection device increases the sperm motility? What are the differences in sperm membrane potential when CA0 is used? Do intracellular Calcium levels change when CA0 is used? Does CA0 increase fertilization rates? Researchers will compare CA0 to the standard of care for sperm selection (density gradient centrifugation) to see if CA0 has similar performance

Participants will:

Provide a semen sample Have their semen sample analyzed, processed and used for assisted reproduction technologies

ELIGIBILITY:
Inclusion Criteria:

* Normozoospermic (18-35 years old) and teratozoospermic (18-60 years old) patients undergoing IVF/ICSI cyles with at least 2 days of sexual abstinence

Exclusion Criteria:

* Less than 4 oocytes collected during oocyte retrieval
* Total sperm count less than 30x10^6

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 115 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-10-30 (Actual); Study Completion 2023-11-15 (Actual)

PRIMARY OUTCOMES:
Sperm membrane potential | Within 2 hours from the sperm collection
  Evaluation of the KCl-induced difference of membrane potential voltage in mV, after sperm selection.
Sperm intracellular Calcium | Within 2 hours from the sperm collection
  Evaluation of the progesterone-induced intracellular calcium fluorescent peaks after sperm selection
Sperm concentration | Within 2 hours from the sperm collection
  Assessment of sperm count after sperm separation
Sperm motility | Within 2 hours from the sperm collection
  Percentage of progresive, non-progressive and immotile sperm after sperm separation
Fertilization rates | 17-20 hours after insemination by IVF or ICSI
  Determination of the rate of 2 pronucleous, 2 polar bodies zygotes after insemination

CONTACTS AND LOCATIONS:
Overall Officials: Claudia L Treviño, Principal Investigator — Departamento de Genética del Desarrollo y Fisiología Molecular, Instituto de Biotecnología (IBT), Universidad Nacional Autónoma de México (UNAM), Cuernavaca, Morelos, México
Locations (1):
- CITMER, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: Yes
Share all IPD that underlie results in the resulting publications
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Starting 12 months after publication of the first resulting publication
Access Criteria: Directly contact investigators

REFERENCES:
- [Background] Allamaneni SS, Agarwal A, Rama S, Ranganathan P, Sharma RK. Comparative study on density gradients and swim-up preparation techniques utilizing neat and cryopreserved spermatozoa. Asian J Androl. 2005 Mar;7(1):86-92. doi: 10.1111/j.1745-7262.2005.00008.x. PMID 15685358
- [Background] Babcock DF. Examination of the intracellular ionic environment and of ionophore action by null point measurements employing the fluorescein chromophore. J Biol Chem. 1983 May 25;258(10):6380-9. PMID 6853488
- [Background] Alpha Scientists in Reproductive Medicine and ESHRE Special Interest Group of Embryology. The Istanbul consensus workshop on embryo assessment: proceedings of an expert meeting. Hum Reprod. 2011 Jun;26(6):1270-83. doi: 10.1093/humrep/der037. Epub 2011 Apr 18. PMID 21502182
- [Background] Brown SG, Publicover SJ, Mansell SA, Lishko PV, Williams HL, Ramalingam M, Wilson SM, Barratt CL, Sutton KA, Da Silva SM. Depolarization of sperm membrane potential is a common feature of men with subfertility and is associated with low fertilization rate at IVF. Hum Reprod. 2016 Jun;31(6):1147-57. doi: 10.1093/humrep/dew056. Epub 2016 Apr 6. PMID 27052499
- [Background] Chen MJ, Bongso A. Comparative evaluation of two density gradient preparations for sperm separation for medically assisted conception. Hum Reprod. 1999 Mar;14(3):759-64. doi: 10.1093/humrep/14.3.759. PMID 10221710
- [Background] Farland LV, Khan SM, Missmer SA, Stern D, Lopez-Ridaura R, Chavarro JE, Catzin-Kuhlmann A, Sanchez-Serrano AP, Rice MS, Lajous M. Accessing medical care for infertility: a study of women in Mexico. F S Rep. 2022 Nov 24;4(1):112-120. doi: 10.1016/j.xfre.2022.11.013. eCollection 2023 Mar. PMID 36959957
- [Background] Henkel RR, Schill WB. Sperm preparation for ART. Reprod Biol Endocrinol. 2003 Nov 14;1:108. doi: 10.1186/1477-7827-1-108. PMID 14617368
- [Background] Hernandez-Silva G, Lopez-Torres AS, Maldonado-Rosas I, Mata-Martinez E, Larrea F, Torres-Flores V, Trevino CL, Chirinos M. Effects of Semen Processing on Sperm Function: Differences between Swim-Up and Density Gradient Centrifugation. World J Mens Health. 2021 Oct;39(4):740-749. doi: 10.5534/wjmh.200115. Epub 2020 Nov 19. PMID 33474848
- [Background] Highland HN, Rishika AS, Almira SS, Kanthi PB. Ficoll-400 density gradient method as an effective sperm preparation technique for assisted reproductive techniques. J Hum Reprod Sci. 2016 Jul-Sep;9(3):194-199. doi: 10.4103/0974-1208.192070. PMID 27803588
- [Background] Hsu CT, Lee CI, Lin FS, Wang FZ, Chang HC, Wang TE, Huang CC, Tsao HM, Lee MS, Agarwal A. Live motile sperm sorting device for enhanced sperm-fertilization competency: comparative analysis with density-gradient centrifugation and microfluidic sperm sorting. J Assist Reprod Genet. 2023 Aug;40(8):1855-1864. doi: 10.1007/s10815-023-02838-4. Epub 2023 Jun 10. PMID 37300647
- [Background] Matamoros-Volante A, Castillo-Viveros V, Torres-Rodriguez P, Trevino MB, Trevino CL. Time-Lapse Flow Cytometry: A Robust Tool to Assess Physiological Parameters Related to the Fertilizing Capability of Human Sperm. Int J Mol Sci. 2020 Dec 24;22(1):93. doi: 10.3390/ijms22010093. PMID 33374265